CLINICAL TRIAL: NCT05839093
Title: Evaluation of the Efficiency of Intraligamentary + Buccal Infiltration Anesthesia and Inferior Alveolar Nerve Block + Buccal Infiltration Anesthesia in Symptomatic Mandibular Molars With Irreversible Pulpitis
Brief Title: Anesthesia Techniques in Symptomatic Mandibular Molars With Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Şehnaz Yilmaz, DDS, PhD, Associated Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDH-2020-12818
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Dental
Keywords: pain; irreversible pulpitis; intraligamentary injection; inferior alveolar nerve block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior Alveolar Nerve Block Group (Active Comparator): A standard Inferior Alveolar Nerve Block (IANB) injection with a conventional dental injector and a 27-G needle to achieve pulpal anesthesia in mandibular molar teeth.
  Interventions: Device: Inferior Alveolar Nerve Block Group
- Intraligamentary Injection Group (Experimental): An intraligamentary injection that performed with a special pressure injection syringe (Sopira Citoject, Kulzer, Hanau, Germany) and a 30-G needle.
  Interventions: Device: Intraligamentary Injection Group

INTERVENTIONS:
Device: Inferior Alveolar Nerve Block Group — A standard IANB injection with a conventional dental injector and a 27-G needle. After determining the injection site and performing aspiration, 1.8 mL of solution was injected at a rate of 1 mL/min to block the inferior alveolar nerve. After achieving lip anesthesia, infiltration was performed at the buccal side of the affected tooth with 0.5 mL using a normal syringe and a 27-G needle. The needle insertion point was the middle of the mesiodistal distance of the crown. Five minutes later, the teeth were isolated and the endodontic procedure was started.
  Arms: Inferior Alveolar Nerve Block Group
Device: Intraligamentary Injection Group — An infiltration was performed at the buccal side of the affected tooth with 0.5 mL using a normal syringe and a 27-G needle. Then, an intraligamentary injection was performed with a special pressure injection syringe (Sopira Citoject, Kulzer, Hanau, Germany) and a 30-G needle. The needle was placed alongside the tooth and inserted at a 30 angle relative to the longitudinal axis of the crown with the needle between the teeth and the bone. Then, in the mesiobuccal, distobuccal, mesiolingual and distolingual portions of teeth, 0.18 mL of the solution was injected. Five minutes later, the teeth were isolated and the endodontic procedure was started.
  Arms: Intraligamentary Injection Group

SUMMARY:
The aim of this clinical study is to evaluate the success of buccal infiltration (BI) anesthesia + intraligamentary (ILI) anesthesia between inferior alveolar nerve block (IANB) anesthesia + buccal infiltration anesthesia in mandibular molar teeth with acute symptomatic irreversible pulpitis.The main questions it aims to answer are:

* Does the anesthesia techniques adequate to perform root canal treatment painlessly?
* Which technique achieved pulpal anesthesia? Participants were allocated in two groups according to the randomization blocks, with a total of 25 patients in each group. In IANB + BI anesthesia techniques, a total of approximately 2.8 ml of anesthetic solution, 1.8 ml + 1 ml, was applied, while for BI + ILI, a total of approximately 1.72 ml, 1 ml + 0.72 ml, was administered. Then, root canal treatment was performed.

Researchers were compared the success of anesthesia techniques in different stages of root canal treatment.

DETAILED DESCRIPTION:
A total of 50 patients, aged between 18-65, who were diagnosed with symptomatic irreversible pulpitis of the mandibular molar tooth, were included in this study. The patients were allocated in two groups according to the randomization blocks, with a total of 25 patients in each group. In IANB + BI anesthesia techniques, a total of approximately 2.8 ml of anesthetic solution, 1.8 ml + 1 ml, was applied, while for BI + ILI, a total of approximately 1.72 ml, 1 ml + 0.72 ml, was administered. After the anesthesia, a rubber dam was placed on the associated tooth of the patient for root canal treatment, the endodontic access cavity was opened, and canal preparation procedures were started. The pain levels felt by the patients during the endodontic treatment stages (starting the treatment, opening the endodontic access cavity and pulp extirpation) were determined by Heft-Parker VAS (HP-VAS) scale. Anesthesia was considered successful in patients who felt no pain (HP-VAS ratio = 0) or mild pain (HP-VAS ratio ≤ 54) during the procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patients
2. The absence of periapical pathology
3. Not sensitive to articaine or epinephrine
4. No facial paresthesia
5. Not taking any analgesic drug 6 hours before treatment
6. Not taking any medication that interferes with anesthesia, such as tricyclic antidepressants and beta-blockers
7. The absence of pathosis in areas planned for injection
8. Not pregnant
9. The absence of pathologic periodontal pockets during probing
10. Patients with a mandibular first molar tooth exhibiting symptomatic irreversible pulpitis

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
The success of anesthesia techniques | 0-2 hours
  Heft-Parker visual analog scale (HPVAS) was used to evaluate the patient's subjective pain and convert it to quantitative values. The pain was classified as follows: 0, no pain as "1"; 1-54 mm, mild pain as "2"; 55-112 mm, moderate pain as "3"; and 114-170 mm, severe pain as "4".
  If the VAS value is 1 and 2, anesthesia is considered successful, if 3 and 4, anesthesia is considered unsuccessful.
  HPVAS-1 determines the VAS value of pain response to cold test. The VAS value of the pain response at the start of the treatment is HPVAS-2.
  The VAS value of the pain response on entering the pulp chamber HPVAS-3:
  The VAS value of the pain response during pulp extirpation was recorded as HPVAS-4.

CONTACTS AND LOCATIONS:
Overall Officials: Şehnaz Yılmaz, DDS,PhD, Principal Investigator — Çukurova University, Faculty of Dentistry
Locations (1):
- Çukurova University, Faculty of Dentistry, Clinic of Endodontics, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It has been collected Visual Analog Scale (VAS) forms from the participants as data. Each participants was marked four times from the beginning to the end of the treatment.
Supporting Information: Study Protocol, SAP
Time Frame: Six months after publication
Access Criteria: Data will be shared only if requested by the editor or referees of the journal that submitted for publication.

REFERENCES:
- [Background] Parirokh M, Yosefi MH, Nakhaee N, Manochehrifar H, Abbott PV, Reza Forghani F. Effect of bupivacaine on postoperative pain for inferior alveolar nerve block anesthesia after single-visit root canal treatment in teeth with irreversible pulpitis. J Endod. 2012 Aug;38(8):1035-9. doi: 10.1016/j.joen.2012.04.012. Epub 2012 May 30. PMID 22794202
- [Background] Habib MFOM, Tarek S, Teama SME, Ezzat K, El Boghdadi RM, Marzouk A, Fouda MY, Gawdat SI, Bedier MM, Amin SAW. Inferior alveolar nerve block success of 2% mepivacaine versus 4% articaine in patients with symptomatic irreversible pulpitis in mandibular molars: A randomized double-blind single-centre clinical trial. Int Endod J. 2022 Nov;55(11):1177-1189. doi: 10.1111/iej.13810. Epub 2022 Aug 20. PMID 35947082

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05839093/Prot_SAP_001.pdf